CLINICAL TRIAL: NCT01689896
Title: Effects of Testosterone Replacement on Pain Sensitivity and Pain Perception in Men With Chronic Pain Syndrome
Brief Title: Testosterone and Pain Sensitivity
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to obtain placebo
Sponsor: Johns Hopkins University (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Adrian S. Dobs, Professor of Medicine and Oncology, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00070640
Record Dates: First submitted 2012-09-11; First posted 2012-09-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Low Testosterone; Hypogonadism; Pain
Keywords: Hypogonadism; Low testosterone; Pain
MeSH Terms: conditions — Hypogonadism; Pain | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone Gel (Active Comparator): Testosterone Gel
  Interventions: Drug: Testosterone Gel
- Placebo Gel (Placebo Comparator): Placebo Gel
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Testosterone Gel
  Other Names: Fortesta®
  Arms: Testosterone Gel
Drug: Placebo Gel
  Arms: Placebo Gel

SUMMARY:
This research is being done to see whether testosterone replacement in men who take opioid-based pain medications and have low testosterone levels will show improvement in pain tolerance, pain perception and quality of life.

Some men who take opioid-based medications (narcotics) for pain develop low testosterone levels. Research has shown that low testosterone levels may make a person more sensitive to pain. This means that if a person with a painful condition develops low testosterone level as a result of his pain medications, he might become more sensitive to pain and so may need higher doses of pain medications for pain control.

Testosterone is a male hormone that is important for sperm production and the development of male characteristics such as muscle mass and strength, fat distribution, bone mass and sex drive. Testosterone hormone replacement therapy has been used for decades to treat men with low testosterone levels (male hypogonadism). Testosterone replacement therapies are available in the form of an injection into the muscle, implants under the skin, oral capsules taken by mouth, topical gels applied to the skin, and skin patches.

This study will use Fortesta®, a topical testosterone gel (T-gel) absorbed into the skin. Fortesta® is currently on the market as an FDA-approved treatment of male hypogonadism (low testosterone levels).

Men with non-cancer related pain who take opioid-based medications for pain and have low testosterone levels may join this study. (A low testosterone level is defined as early morning (before noon) blood testosterone level of 300 ng/dl or less, or a free testosterone of 50 ng/dl or less)).

ELIGIBILITY:
Inclusion Criteria:

* Men
* 18 Years of Age and Older
* Serum total testosterone level <300 ng/dl or free testosterone < 50 pg/ml
* Consumption of at least 10 mg of hydrocodone (or analgesic equivalent of another opioid) for at least 4 weeks
* Absence of hospitalization in past 2 months
* No acute illness in past 2 months
* No prior history of any form of hypogonadism
* No current anabolic therapy (growth hormone, DHEA, etc)
* No current use or consumption in past 2 months of glucocorticoids and melatonin
* Normal digital rectal examination
* Normal PSA level

Exclusion Criteria:

* Liver enzymes >3 times upper limit of normal
* Serum creatinine > 2 times upper limit of normal
* Neurological disease
* Active psychiatric illness
* Any addictive and/or illicit drug use
* Alcoholism (>10 drinks/week)
* Patients currently receiving glucocorticoids, melatonin or anabolic agents
* Hospitalization in past 2 months
* Acute illness in past 2 months
* Consumption of < 20 mg of hydrocodone (or analgesic equivalent of another opioid)
* Severe BPH
* PSA >4.0 ng/ml
* Prostate cancer
* Breast cancer
* Any cancer or cancer related pain
* History of alcohol abuse
* Known peripheral neuropathy (any etiology) or peripheral vascular disease (including Raynaud's disease), which may interfere with pain testing
* Concurrent warfarin treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain Tolerance - CPT | 18 weeks
  Cold Pressor Test: Participants will undergo a standard cold pressor task consisting of immersion of the right hand in a 4°C circulating water bath. The standardized instructions for the procedure will direct participants to keep their hands in the water for as long as possible but if the sensations become intolerable participants can remove their hands at any time. At the conclusion of the trial, participants will provide 0-100 ratings of the maximum intensity and unpleasantness of pain produced by water immersion during the trial. During the immersion trial, the time to cold pain threshold (CPTH), pain intensity and tolerance (CPTO) will be recorded.
Pain Tolerance - PPT | 18 Weeks
  Pressure Pain Test: A Somedic algometer will be used to assess responses to noxious mechanical pressure. Pressure is increased steadily at a constant rate until the subject responds by pressing a button, at which point stimulation is terminated. Pressure pain thresholds and tolerances will be assessed 2 times each at 3 body sites bilaterally (the order of which will be randomized): trapezius muscle, masseter muscle, biceps femoris muscle, and ulnar area. For trials of pressure pain threshold, subjects indicate when the stimulus "first feels painful" and for trials of pressure pain tolerance, subjects are asked to respond when the stimulus "becomes intolerable."
QOL | 18 Weeks
  Quality of Life: This parameter will be evaluated using Short Form-36 (SF-36) questionnaire.
Pain Tolerance - TPPT | 18 Weeks
  Thermal Pain Perception Test: Contact heat stimuli will be delivered using a Medoc Thermal Sensory Analyzer, a peltier-element-based stimulator, with the 9 cm2 contact probe applied to the left forearm. The initial thermal assessment procedures include sampling of heat pain thresholds and heat pain tolerances using an ascending method of limits paradigm with a rate of rise of .5°C /Sec.
  Following, a series of 3 temporal summation procedures will be administered. Sequences of 10 rapid heat pulses are to be applied to the left volar forearm. Target temperatures will be based on subjects' individualized pain thresholds. Subjects will verbally rate the painfulness of each thermal pulse on a 0-100 (0= "no pain", 100= "most intense pain imaginable") rating scale. Subjects will be able to terminate the procedure at any time; for those who do, value equivalents to the final rating preceding termination will be assigned to the remaining trials for statistical analysis.

SECONDARY OUTCOMES:
Hormonal Outcomes | 18 Weeks
  Serum will be obtained for serum total and free testosterone, estradiol, prolactin, SHBG, DHEA, FSH, and LH. Bone markers in the form of spot urine N-telopeptides, bone-specific alkaline phosphatase and osteocalcin will be checked, as a measure of bone turnover.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States